CLINICAL TRIAL: NCT01772303
Title: An Open-Label, Prospective, Multicenter Study to Assess the Safety and Efficacy of HO/03/03 10-40 Micro Gram (Wound Size Dependence) Applied Topically for up to 24 Weeks in Subjects With Various Etiologies of Hard-to-Heal Wounds
Brief Title: Safety and Efficacy Study of HO/03/03 10-40 Micro Grams to Treat Hard to Heal Wounds
Acronym: H2H
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HealOr (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO-H2H-01-2011
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Hard to Heal Wounds
Keywords: Pressure Ulcers, diabetic Ulcers, post operational wounds
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HO/03/03 10-40 micro gram (Experimental): Topically treatment with HO/03/03 10-40µg once daily for up to 24 weeks. Subjects will receive treatment with HO/03/03 10µg at a dose of 1-4 vials (i.e. 10-40 µg/administration) daily depending on their wound size.
  Interventions: Drug: HO/03/03 10-40 µg

INTERVENTIONS:
Drug: HO/03/03 10-40 µg — HO/03/03 10-40µg once daily (Topically) for up to 24 weeks.

SUMMARY:
This multicenter, prospective, open-label, outpatient study will assess the safety and efficacy of HO/03/03 10µg applied topically once daily for up to 24 weeks in up to 100 subjects with Hard to Heal documented chronic wounds of various etiologies (pressure ulcers, diabetic ulcers, post operational wounds surgical incisions ulcers of rheumatoid arthritis and trauma wounds) of at least 4 weeks documentation.

DETAILED DESCRIPTION:
All subjects with a wound size of up to 56.25 cm2 (inclusive) will be administered 1 vial of 10 ml HO/03/03 10μg per administration. For each increase in wound size of up to 56.25 cm2 an additional vial of HO/03/03 10 μg will be added up to a maximal wound size area of 225 cm2 (will be measured by HealOr central reviewer) utilizing 40µg (4 vials) per administration. 15 min post treatment wounds will be dressed according to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old and above.
* Chronic wounds that have < 30% change in area from Screening
* Have single / multiple wounds;
* Have a Hard-to-Heal wound(s) of various etiologies

Exclusion Criteria:

* Have a documented medical history of a significant cardiac, pulmonary, gastrointestinal, endocrine (other than Diabetes Mellitus type 1 or 2), hepatic or per the physician's discretion.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Time to Heal | up to 24 weeks
  1. 75% wound closure by or on study week 24 (Time to Event Analysis of incidence and time to 75% wound closure).

SECONDARY OUTCOMES:
Wound closure | up to 24 weeks
  1. Complete wound closure by or on week 24 (Time to Event Analysis of incidence and time to 100% wound closure).

CONTACTS AND LOCATIONS:
Locations (1):
- Maccabi Health Services, Wound Clinic, Haifa, Israel